CLINICAL TRIAL: NCT06670872
Title: A Study on the Combination Therapy of Eravacycline for Treating Carbapenem-Resistant Acinetobacter Baumannii Pneumonia
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, WangFei, chief physician, Peking University Third Hospital
Other Study IDs: M2024219
Record Dates: First submitted 2024-10-21; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Pneumonitis; Acinetobacter Baumannii
Keywords: Eravacycline
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Eravacycline combination therapy group: Eravacycline is administered intravenously at a dosage of 1mg/kg, once every 12 hours. The duration of intravenous infusion is approximately 60 minutes.The combined drugs include sulbactam or compound preparations containing sulbactam, polymyxin B, beta-lactam antibiotics, etc., used according to their instructions for use or clinical practice guidelines.
  Interventions: Drug: Eravacycline combination therapy group

INTERVENTIONS:
Drug: Eravacycline combination therapy group — Physicians determine the combination regimen of eravacycline, which may include sulbactam or compound preparations containing sulbactam, polymyxin B, beta-lactam antibiotics, etc., based on the pathogen identification and susceptibility results, and the China Guidelines for Diagnosis, Treatment, and Prevention of Infections Caused by Carbapenem-Resistant Gram-Negative Bacteria." The combined drugs are used according to their instructions for use or clinical practice guidelines.

SUMMARY:
This study intends to evaluate the efficacy and safety of eravacycline-based combination therapy in real words for Chinese patients with CRAB pneumonia, providing data reference for clinical treatment of CRAB pneumonia.

DETAILED DESCRIPTION:
This study aims to include 50 patients proven or suspected diagnosed carbapenem-resistant Acinetobacter baumannii pneumonia at Peking University Third Hospital. The physician determines to use a combination regimen of eravacycline, including sulbactam or compound preparations containing sulbactam, polymyxin B, and β-lactam antibiotics, is considered. The clinical response rate at the end of treatment is the primary endpoint of the study; the secondary endpoints include the clearance rate of carbapenem-resistant Acinetobacter baumannii, the incidence of adverse events, and the all-cause mortality rate within 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Voluntarily participating in this study and signing an informed consent form. If the subject is unable to read and/or sign the informed consent form due to lack of capacity or other reasons, the informed process and the informed consent form must be signed by their legal guardian.
3. Patients with clinical manifestations and imaging results consistent with bacterial pneumonia, and who are expected to benefit from antimicrobial treatment. Suspected carbapenem-resistant Acinetobacter baumannii infection or Acinetobacter baumannii detected in two consecutive sputum cultures (at least one of which must be from bronchoalveolar lavage or endotracheal aspirate), with resistance to carbapenems.
4. Patients who have been treated with eravacycline for at least 3 days.

Exclusion Criteria:

1. The investigator believes that there are any medical history, current condition, treatment, abnormal laboratory test results, or other situations that may affect the trial results, interrupt the trial process (or the subject cannot complete all trial requirements, operations, and visits), or increase the risk to the subject from receiving the trial medication, including patients with terminal illness, or evidence of an immediately life-threatening disease.
2. Patients with a history of allergic reactions to tetracyclines or any excipients contained in the formulation of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study plans to include patients proven or suspected diagnosed of carbapenem-resistant Acinetobacter baumannii pneumonia, who are 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
clinical efficacy at the end of treatment | up to the end of treatment, up to 4 weeks(estimation)
  The primary endpoint is the clinical efficacy at the end of treatment (within 24 hours after the last dose of the trial medication) for all patients who have completed the trial according to the protocol. Clinical efficacy is assessed and the clinical response rate is calculated.
  Clinical response is evaluated by PI，and defined as an improvement, reduction, or disappearance of the patient's multiple symptoms and signs compared to before treatment, along with improvement or normalization of imaging findings.
  Clinical response rate = (number of patients with symptom relief) / (total number of patients included in the study).

SECONDARY OUTCOMES:
Incidence Rate of Adverse Event | up to the end of treatment, up to 4 weeks(estimation)
  safety data according to CTC-AE
The microbiological clearance rate | up to the end of treatment, up to 4 weeks(estimation)
  The microbiological clearance rate is at the end of treatment
The all cause mortality rate | 28 days
  The all-cause mortality rate within 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Wang Fei, doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China